CLINICAL TRIAL: NCT03553862
Title: The Impact of Collaborative Care Model in the Management of Primary Care Patients With Type 2 Diabetes Mellitus in Singapore
Brief Title: Collaborative Care Model on Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Joyce Lee, PharmD, Principle Investigator, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017/01191
Record Dates: First submitted 2018-05-09; First posted 2018-06-12 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients randomly assigned to the control arm will receive the usual or conventional care not interfered by the study team.
- Intervention (Experimental): The intervention arm will receive collaborative care from a team of healthcare professionals that consists of pharmacist, physicians, nurses and dietitians. Patients in the intervention group will also receive clinical interventions carried out by the pharmacist.
  Interventions: Behavioral: collaborative care

INTERVENTIONS:
Behavioral: collaborative care — The intervention arm will receive collaborative care from a team of healthcare professionals that consists of pharmacist, physicians, nurses and dietitians. Patients in the intervention group will also receive clinical interventions carried out by the pharmacist.nurses and dietitians as well as a pharmacist.
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine the effectiveness of the collaborative care model in Singapore in which clinical pharmacists, nurses and dietitians are active participants who collaborate with physicians in caring for patients with Type 2 diabetes mellitus (DM).Since DM is a cardiovascular risk equivalent, co-morbidities such as hypertension (HTN) and dyslipidaemia (DLP) will also be evaluated to assess the holistic care provided for the investigator's patients afflicted with these top chronic diseases in Singapore.

DETAILED DESCRIPTION:
Specifically, this study aims to evaluate the effectiveness of an integrated collaborative care model comprising of a healthcare team (physician, clinical pharmacist, nurse, and/or dietitian) compared to the usual or conventional healthcare model (physician-centered care) mainly in the clinical, humanistic and economic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 21 years with Type 2 DM (HbA1c > 7%) and polypharmacy (≥ 5 medications) will be eligible for this study.

Exclusion Criteria:

* Patients with Type 1 DM or who are unable to communicate independently in English, Chinese or Malay will be excluded from this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline Body mass index (BMI) at 6-month | baseline and 6-month
  Change of BMI in kg/m^2
Change from baseline Glycated Haemoglobin (HbA1c) at 6-month | baseline and 6-month
  Change of HbA1c in %
Changes from baseline Systolic Blood Pressure (SBP) at 6-month | baseline and 6-month
  Change of SBP in mmHg
Change from baseline Low-density lipoprotein (LDL) at 6-month | baseline and 6-month
  Change of LDL in mg/dL
Change from baseline High-density lipoprotein (HDL) at 6-month | baseline and 6-month
  Change of HDL in mg/dL
Change from baseline Total cholesterol (TC) at 6-month | baseline and 6-month
  Change of TC in mg/dL
Change from baseline Glycerides (TG) at 6-month | baseline and 6-month
  Changes of TG in mg/dL
Incidence of hypoglycaemia | 6-month
  Incidence of hypoglycaemia
Change from baseline Body mass index (BMI) at 12 months | 12-month
  Change BMI in kg/m^2
Change from baseline Glycated Haemoglobin (HbA1c) at 12-month | 12-month
  Changes of HbA1c in %
Change from baseline Systolic Blood Pressure (SBP) at 12-month | 12-month
  Change of SBP in mmHg
Change from baseline Low-density lipoprotein (LDL) at 12-month | 12-month
  Changes of LDL in mg/dL
Change from baseline High-density lipoprotein (HDL) at 12-month | 12-month
  Changes of HDL in mg/dL
Change from baseline Total cholesterol (TC) at 12-month | 12-month
  Changes of TC in mg/dL
Change from baseline Glycerides (TG) at 12-month | 12-month
  Changes of TG in mg/dL
Incidence of hypoglycaemia | 12-month
  Incidence of hypoglycaemia

SECONDARY OUTCOMES:
The 5-level EQ-5D version (5Q-5D-5L) | baseline
  5Q-5D-5L is a questionnaire containing 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) with 5 levels (no problems, slight problems, moderate problems, severe problems and extreme problems) for the patients to indicate their health stage.
The 5-level EQ-5D version (5Q-5D-5L) | 6-month
  5Q-5D-5L is a questionnaire containing 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) with 5 levels (no problems, slight problems, moderate problems, severe problems and extreme problems) for the patients to indicate their health stage.
The 5-level EQ-5D version (5Q-5D-5L) | 12-month
  5Q-5D-5L is a questionnaire containing 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) with 5 levels (no problems, slight problems, moderate problems, severe problems and extreme problems) for the patients to indicate their health stage.
Audit of Diabetes Dependent Quality of Life (ADDQoL) | baseline
  The ADDQoL is a 19-item questionnaire measuring the effects of diabetes and its treatment on individuals' quality of life.
Audit of Diabetes Dependent Quality of Life (ADDQoL) | 6-month
  The ADDQoL is a 19-item questionnaire measuring the effects of diabetes and its treatment on individuals' quality of life.
Audit of Diabetes Dependent Quality of Life (ADDQoL) | 12-month
  The ADDQoL is a 19-item questionnaire measuring the effects of diabetes and its treatment on individuals' quality of life.
The Problem Area in Diabetes (PAID) | baseline
  The PAID is a valid and reliable 20-item questionnaire measuring diabetes-related distress with a five-point Likert scale that ranges from 0 (not a problem) to 4 (serious problem).
The Problem Area in Diabetes (PAID) | 6-month
  The PAID is a valid and reliable 20-item questionnaire measuring diabetes-related distress with a five-point Likert scale that ranges from 0 (not a problem) to 4 (serious problem).
The Problem Area in Diabetes (PAID) | 12-month
  The PAID is a valid and reliable 20-item questionnaire measuring diabetes-related distress with a five-point Likert scale that ranges from 0 (not a problem) to 4 (serious problem).
Summary of Diabetes Self-Care Activities (SDSCA) | baseline
  The SDSCA measure is a brief self-report questionnaire of diabetes self-management that includes 14 items assessing the following aspects of the diabetes regimen: general dies, specific diet, exercise, blood-glucose testing, foot care, and smoking.
Summary of Diabetes Self-Care Activities (SDSCA) | 6-month
  The SDSCA measure is a brief self-report questionnaire of diabetes self-management that includes 14 items assessing the following aspects of the diabetes regimen: general dies, specific diet, exercise, blood-glucose testing, foot care, and smoking.
Summary of Diabetes Self-Care Activities (SDSCA) | 12-month
  The SDSCA measure is a brief self-report questionnaire of diabetes self-management that includes 14 items assessing the following aspects of the diabetes regimen: general dies, specific diet, exercise, blood-glucose testing, foot care, and smoking.
Self-report Hypoglycaemia Question | baseline
  It is 5-item questionnaire for the patients with diabetes to self-assess their symptoms of hypoglycaemia.
Self-report Hypoglycaemia Question | 6-month
  It is 5-item questionnaire for the patients with diabetes to self-assess their symptoms of hypoglycaemia.
Self-report Hypoglycaemia Question | 12-month
  It is 5-item questionnaire for the patients with diabetes to self-assess their symptoms of hypoglycaemia.
Work Productivity and Activity Impairment questionnaire, General Health version (WPAI-GH) | 6-month
  The WPAI-GH is a 6-item questionnaire measuring absenteeism, presenteeism, overall work productivity loss, and daily activity impairment with a 10-point scale that range from 0 (no effect on daily activities) to 10 (serious effect on daily activities).
Work Productivity and Activity Impairment questionnaire, General Health version (WPAI-GH) | 12-month
  The WPAI-GH is a 6-item questionnaire measuring absenteeism, presenteeism, overall work productivity loss, and daily activity impairment with a 10-point scale that range from 0 (no effect on daily activities) to 10 (serious effect on daily activities).

CONTACTS AND LOCATIONS:
Overall Officials: Wei Yan Tan, Principal Investigator — National Healthcare Group Pharmacy
Locations (1):
- Chua Chu Kang Polyclinic, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siaw MYL, Ko Y, Malone DC, Tsou KYK, Lew YJ, Foo D, Tan E, Chan SC, Chia A, Sinaram SS, Goh KC, Lee JY. Impact of pharmacist-involved collaborative care on the clinical, humanistic and cost outcomes of high-risk patients with type 2 diabetes (IMPACT): a randomized controlled trial. J Clin Pharm Ther. 2017 Aug;42(4):475-482. doi: 10.1111/jcpt.12536. Epub 2017 Apr 27. PMID 28449205
- [Background] Jarab AS, Alqudah SG, Mukattash TL, Shattat G, Al-Qirim T. Randomized controlled trial of clinical pharmacy management of patients with type 2 diabetes in an outpatient diabetes clinic in Jordan. J Manag Care Pharm. 2012 Sep;18(7):516-26. doi: 10.18553/jmcp.2012.18.7.516. PMID 22971205
- [Background] Scott DM, Boyd ST, Stephan M, Augustine SC, Reardon TP. Outcomes of pharmacist-managed diabetes care services in a community health center. Am J Health Syst Pharm. 2006 Nov 1;63(21):2116-22. doi: 10.2146/ajhp060040. PMID 17057049
- [Background] Taylor KI, Oberle KM, Crutcher RA, Norton PG. Promoting health in type 2 diabetes: nurse-physician collaboration in primary care. Biol Res Nurs. 2005 Jan;6(3):207-15. doi: 10.1177/1099800404272223. PMID 15583361

DOCUMENTS (1):
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT03553862/Prot_000.pdf